CLINICAL TRIAL: NCT02882594
Title: Testing the Reliability and Validity of the CIBA
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-2812
Record Dates: First submitted 2016-08-15; First posted 2016-08-30 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Quality Improvement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- CIBA Study Cohort: Patients aged 1 to 13 years undergoing inhalation inductions for general anesthesia
  Interventions: Behavioral: Observing patient behaviors for anesthesia induction compliance

INTERVENTIONS:
Behavioral: Observing patient behaviors for anesthesia induction compliance — Observing patient behaviors for anesthesia induction compliance so to test reliability and validity of the CIBA Tool

SUMMARY:
The overall objective of the study is to improve the experience for pediatric patients undergoing anesthesia inductions. The specific objective for this proposal is to establish whether the CIBA tool demonstrates inter-rater reliability and concurrent validity with the Induction Compliance Checklist.

DETAILED DESCRIPTION:
The proposed research study will assess the reliability and validity of a new tool that is being used in the Department of Anesthesia (The Child Induction Behavioral Assessment tool) to grade the difficulty of patient behaviors exhibited during anesthesia inductions. The Child Induction Behavioral Assessment (CIBA) tool is more succinct than previously validated tools for assessing behavioral responses to inhalation inductions, making it practical for use in a busy clinical practice setting. Having clinicians document a patient's behavioral response to induction using the CIBA tool is useful because this information can help to optimize subsequent induction plans if the patient returns. Additionally, population data may be collected using electronic data reports for QI purposes. Prior to using data from the CIBA tool in QI initiatives, it is important to assess whether this tool is reliable and valid.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to Same Day Surgery department at CCHMC base campus for any surgical or Intervention Radiology procedure
* Ages 1-13 years old
* Male or female
* Patients of any ethnicity
* Family and participant communicate primarily in English
* Patients with normal neurocognitive development
* Patients undergoing inhalation induction using an anesthesia mask
* American Society of Anesthesiologists (ASA) physical classification status I, II, or III
* Patients who do or do not receive a premedication for anxiety
* Parent/guardian present at the induction of anesthesia

Exclusion Criteria:

* Guardian unavailable to give consent
* Neurocognitive delays
* Tracheostomy
* Intravenous (IV) induction or nitrous sedation prior to IV induction
* Coordinators unable to observe or fully observe the induction
* CIBA assessment not completed by anesthesia provider

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: patients aged 1 to 13 years undergoing inhalation inductions for general anesthesia
Sampling Method: Probability Sample
Enrollment: 384 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Test the reliability and validity of the Child Induction Behavioral Assessment (CIBA) Tool by evaluating inter-rater reliability and concurrent reliability and validity of the CIBA tool with the already validated Induction Compliance Checklist (ICC) | two years

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Winterberg AV, Ding L, Hill LM, Stubbeman BL, Varughese AM. Validation of a Simple Tool for Electronic Documentation of Behavioral Responses to Anesthesia Induction. Anesth Analg. 2020 Feb;130(2):472-479. doi: 10.1213/ANE.0000000000003945. PMID 30531219